CLINICAL TRIAL: NCT05588336
Title: Comparison of the Effects of Intrathecal Morphine at Two Different Doses in Thoracoscopic Lung Resection
Brief Title: Intrathecal Morphine for Thoracoscopic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, associate professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ITM1
Record Dates: First submitted 2022-10-12; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
Keywords: postoperative analgesia; pain score; side effect; morphine; intrathecal
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 mcg/kg intrathecal morphine (Active Comparator): For postoperative analgesia, before surgical incision, 10 mcg/ideal body weight morphine HCl (in 2 ml volume) was administered intrathecally at L4-5 interspace in the lateral decubitis position.
  Interventions: Drug: Morphine
- 7 mcg/kg intrathecal morphine (Active Comparator): For postoperative analgesia, before surgical incision 7 mcg/ideal body weight morphine HCl (in 2 ml volume) was administered intrathecally at L4-5 interspace in the lateral decubitis position.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — In the literature, intrathecal morphine doses were applied according to the patients' actual body weight and there is no study comparing intrathecal morphine dose in thoracic surgery patients.

SUMMARY:
Thoracic surgery is one of the surgeries where postoperative pain is intense. In this study, the investigators aimed to compare the efficacy of two different intrathecal morphine doses administered for postoperative analgesia according to patients' ideal body weight.

DETAILED DESCRIPTION:
Patients who underwent video-assisted thoracic surgery were divided into two groups: 10 mcg/kg and 7 mcg/kg intrathecal morphine for postoperative analgesia. Intraoperative and postoperative hemodynamic variables, postoperative morphine consumption, postoperative pain scores, side effects and additional analgesic requiretment were recorded.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* ASA class I and II
* Video-assisted thoracoscopic surgery

Exclusion Criteria:

* < 18 years old
* ASA class > II
* Serious hepatic, cardiac, renal, metabolic, endocrine diseases
* Coagulation disfunction
* Allergy to any of the study drugs
* Pneumonectomy
* Infection in the lumbar region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
pain scores | Change from baseline pain scores at 24 hours
  Postoperative pain scores of the patients were recorded via Visual Analog Scale (VAS; 0= no pain, 10= worst pain)
morphine consumption | Change from baseline morphine consumption at 24 hours
  At the end of surgery, patients were allowed to use the patient controlled analgesia (PCA) device. The PCA delivered bolus doses of morphine (0.02 mg/kg) every 10 minutes without a backround infusion. Morphine consumption (mg) was evaluated and recorded postoperative 24 hours.

SECONDARY OUTCOMES:
systolic arterial blood pressure | change from baseline systolic blood pressure at 150 minutes
  Intraoperative systolic arterial blood pressure (mmHg) values were recorded during surgery.
diastolic arterial blood pressure | change from baseline diastolic blood pressure at 150 minutes
  Intraoperative diastolic arterial blood pressure (mmHg) values were recorded during surgery.
mean arterial blood pressure | change from baseline mean arterial blood pressure at 150 minutes
  Intraoperative mean arterial blood pressure (mmHg) values were recorded during surgery.
heart rate | change from baseline heart rate at 150 minutes
  Intraoperative heart rate (beats/minute) values were recorded during surgery.
side effects | postoperative 24 hours
  All of patients were visited in the thoracic surgery ward after surgery and side effects were evaluated and recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)